CLINICAL TRIAL: NCT03648645
Title: Hypertensive Pregnant Women Monitored by Teletransmitted Self-measurements of Blood Pressure
Acronym: FETH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 35RC17_8837_FETH
Record Dates: First submitted 2018-08-21; First posted 2018-08-27 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Hypertension in Pregnancy
Keywords: Pregnancy; Hypertension; telemonitoring
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AH Telemonitoring (Experimental): Self measurement of blood pressure
  Interventions: Device: Self measurement of blood pressure

INTERVENTIONS:
Device: Self measurement of blood pressure — Patients will perform the measurement of blood pressure at home, on a daily basis, in complying with the "rule of 3" stated by the Haute Autorité de Santé (French Health Authority) : i.e. 3 consecutive measurements in the morning and in the evening, after a period of rest Measurements are performed using a blood pressure monitor Bluetooth-connected. If a threshold value is exceeded (and depending on the alert), a consultation will be scheduled (unexpected consultation) and notified to the patient.

SUMMARY:
The occurrence of arterial hypertension (AH) during pregnancy is a major cause of fetal, neonatal and maternal morbidity and mortality in western countries. It is estimated that about 10% of pregnancies are complicated by AH (80 000 women / year in France). It is therefore essential to diagnose AH with certainty in order to set-up appropriate care and follow its evolution.

DETAILED DESCRIPTION:
The objective of this study is to show the faisability of self-measurement with teletransmission for long-term follow-up of hypertensive pregnant women (at high risk of preeclampsia) by avoiding repeated, prolonged visits or hospitalizations and to optimize the intervention of health professionals by providing them with reliable data.

A multicenter, controlled study will be conducted in women presenting with mild to moderate hypertension without preeclampsia followed throughout their pregnancy by either self-measurement with teletransmission.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with confirmed mild to moderate AH untreated and / or under antihypertensive treatment (for gestational or chronic hypertension)
* Women without preeclampsia requiring enhanced AH surveillance
* Patient affiliated to a social security system
* Patient giving consent to participate in the study.
* Age> 18 years

Exclusion Criteria:

* arm circumference greater than 42 cm unsuitable for self-measurement,
* women in atrial fibrillation, or frequently in arrhythmia, with secondary hypertension or severe hypertension or with cardiovascular complication.
* women having preeclampsia.
* women having an AH by "white coat effect".
* women having a move or maternity change planned during pregnancy.
* majors protected under tutorship or curatorship, or under the protection of justice.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Hypertension specific intervention | Through study completion, an average of 9 months
  Percentage of blood pressure measurements initially planned and actually performed during the course of the investigation

SECONDARY OUTCOMES:
Number of blood pressure measurements per day and per week | Through study completion, an average of 9 months
Likert scale to assess patients' satisfaction | Through study completion, an average of 9 months
  Evaluation of the patients' satisfaction regarding their medical care during pregnancy assessed by Likert scale : from 1 (Very dissatisfied) to 5 (Very satisfied)
Likert scale to assess medical staff's satisfaction | Through study completion, an average of 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Thierry DENOLLE, MD, Study Director — Hospital of Dinard
Locations (5):
- France (5):
  - CHU Caen, Caen
  - CHU Lille, Lille
  - Hôpital Cochin (APHP), Paris
  - CH St-Malo, St-Malo
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ashworth DC, Maule SP, Stewart F, Nathan HL, Shennan AH, Chappell LC. Setting and techniques for monitoring blood pressure during pregnancy. Cochrane Database Syst Rev. 2020 Jul 23;8(8):CD012739. doi: 10.1002/14651858.CD012739.pub2. PMID 32748394